CLINICAL TRIAL: NCT00963599
Title: A Multicenter, Double-Blind, Randomized, Parallel-Group Study Investigating the Clinical Effect of Combination Montelukast/Loratadine in Patients With Seasonal Allergic Rhinitis-Fall Study
Brief Title: Montelukast in Seasonal Allergic Rhinitis - Fall 1999 Study (0476A-117)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0476A-117; MK0476A-117; 2009_645
Record Dates: First submitted 2009-08-19; First posted 2009-08-21 (Estimated); Results first posted 2010-06-16 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Loratadine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Experimental): montelukast/loratadine
  Interventions: Drug: Comparator: montelukast/loratadine
- 2 (Experimental): loratadine
  Interventions: Drug: Comparator: loratadine
- 3 (Experimental): montelukast
  Interventions: Drug: Comparator: montelukast
- 4 (Placebo Comparator): placebo
  Interventions: Drug: Comparator: placebo

INTERVENTIONS:
Drug: Comparator: montelukast/loratadine — montelukast 10 mg/loratadine 10 mg tablet taken once daily at bed time for 2 weeks
  Arms: 1
Drug: Comparator: montelukast — montelukast 10 mg tablet taken once daily at bed time for 2 weeks
  Arms: 3
Drug: Comparator: loratadine — loratadine 10 mg tablet taken once daily at bed time for 2 weeks
  Arms: 2
Drug: Comparator: placebo — placebo tablet taken once daily at bed time for 2 weeks
  Arms: 4

SUMMARY:
This study will evaluate the ability of oral montelukast/loratadine to improve the signs and symptoms of seasonal allergic rhinitis compared with loratadine alone, montelukast alone and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a documented history of seasonal allergic rhinitis symptoms that flare up during the study season
* Patient is a nonsmoker
* Patient is in good general health

Exclusion Criteria:

* Patient is hospitalized
* Patient is a woman who is less than 8 weeks postpartum or is breast-feeding
* Patient intends to move or vacation away during the study
* Patient has had any major surgery within 4 weeks of study start
* Patient is a current or past abuser of alcohol or illicit drugs
* Patient has been treated in an emergency room for asthma in the past month
* Patient had an upper respiratory infection with in 3 weeks prior to study start
* Patient has any active pulmonary disorder other than asthma

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 907 (Actual)
Dates: Start 1999-09; Primary Completion 1999-11 (Actual); Study Completion 1999-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Nayak AS, Philip G, Lu S, Malice MP, Reiss TF; Montelukast Fall Rhinitis Investigator Group. Efficacy and tolerability of montelukast alone or in combination with loratadine in seasonal allergic rhinitis: a multicenter, randomized, double-blind, placebo-controlled trial performed in the fall. Ann Allergy Asthma Immunol. 2002 Jun;88(6):592-600. doi: 10.1016/S1081-1206(10)61891-1. PMID 12086367

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty study centers in the United States.
  Therapy Period: September 1999 to November 1999
Pre-assignment Details: Patients who required excluded medication and those who did not meet a minimum predefined level of combined Daytime Nasal Symptoms score during the run-in period were excluded from randomization.
Groups:
- Placebo: Matching-image placebo tablet to each of montelukast, loratadine, and montelukast/loratadine combination orally once daily at bedtime for 2 weeks
- Montelukast: Montelukast 10 mg tablet and matching-image placebo tablet to each of loratadine and montelukast/loratadine combination orally once daily at bedtime for 2 weeks
- Loratadine: Loratadine 10 mg tablet and matching-image placebo tablet to each of montelukast and montelukast/loratadine combination orally once daily at bedtime for 2 weeks
- Montelukast/Loratadine: Montelukast 10 mg/loratadine 10 mg combination tablet and matching-image placebo tablet to each of montelukast and loratadine orally once daily at bedtime for 2 weeks
Period: Overall Study
Arm/Group | Placebo | Montelukast | Loratadine | Montelukast/Loratadine
Started | 149 | 155 | 301 | 302
Completed | 143 | 149 | 292 | 288
Not Completed | 6 | 6 | 9 | 14
Not completed — Adverse Event | 2 | 0 | 1 | 2
Not completed — Lack of Efficacy | 0 | 2 | 1 | 4
Not completed — Lost to Follow-up | 0 | 1 | 1 | 1
Not completed — Protocol Violation | 2 | 2 | 3 | 4
Not completed — Withdrawal by Subject | 2 | 1 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Montelukast | Loratadine | Montelukast/Loratadine | Total
Number analyzed (Participants) | 149 | 155 | 301 | 302 | 907
Age, Continuous [Mean (Full Range); unit: Years] | 36.9 [15 to 81] | 35.2 [15 to 65] | 37.1 [15 to 82] | 37.6 [15 to 78] | 36.9 [15 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 102 | 191 | 208 | 587
  Male | 63 | 53 | 110 | 94 | 320
Composite Symptoms Score (Daytime Nasal and Nighttime Symptoms) [Mean (Standard Deviation); unit: Units on a Scale] — 0 (best) to 3 (worst) point scale
  Units on a Scale | 1.71 (0.45) | 1.82 (0.43) | 1.82 (0.45) | 1.78 (0.46) | 1.79 (0.45)
Daytime Congestion score [Mean (Standard Deviation); unit: Units on a Scale] — 0 (best) to 3 (worst) point scale
  Units on a Scale | 2.26 (0.56) | 2.31 (0.50) | 2.37 (0.52) | 2.31 (0.58) | 2.32 (0.54)
Daytime Eye Symptoms Score [Mean (Standard Deviation); unit: Units on a Scale] — 0 (best) to 3 (worst) point scale
  Units on a Scale | 1.31 (0.73) | 1.38 (0.73) | 1.38 (0.78) | 1.38 (0.77) | 1.37 (0.76)
Daytime Nasal Itching score [Mean (Standard Deviation); unit: Units on a Scale] — 0 (best) to 3 (worst) point scale
  Units on a Scale | 1.94 (0.67) | 1.94 (0.70) | 1.93 (0.79) | 1.89 (0.73) | 1.92 (0.74)
Daytime Nasal Symptoms Score [Mean (Standard Deviation); unit: Units on a Scale] — 0 (best) to 3 (worst) point scale
  Units on a Scale | 2.01 (0.44) | 2.06 (0.39) | 2.09 (0.44) | 2.01 (0.43) | 2.04 (0.43)
Daytime Rhinorrhea score [Mean (Standard Deviation); unit: Units on a Scale] — 0 (best) to 3 (worst) point scale
  Units on a Scale | 2.02 (0.70) | 2.05 (0.61) | 2.16 (0.58) | 1.98 (0.66) | 2.06 (0.64)
Daytime Sneezing score [Mean (Standard Deviation); unit: Units on a Scale] — 0 (best) to 3 (worst) point scale
  Units on a Scale | 1.81 (0.74) | 1.93 (0.65) | 1.89 (0.74) | 1.87 (0.68) | 1.87 (0.71)
Nasal Congestion Upon Awakening [Mean (Standard Deviation); unit: Units on a Scale] — 0 (best) to 3 (worst) point scale
  Units on a Scale | 2.17 (0.65) | 2.25 (0.56) | 2.26 (0.61) | 2.20 (0.63) | 2.23 (0.62)
Nighttime Symptoms Score [Mean (Standard Deviation); unit: Units on a Scale] — 0 (best) to 3 (worst) point scale
  Units on a Scale | 1.32 (0.65) | 1.50 (0.64) | 1.47 (0.63) | 1.46 (0.66) | 1.45 (0.65)
Rhinoconjunctivitis Quality-of-Life Score [Mean (Standard Deviation); unit: Units on a Scale] — 0 (best) to 6 (worst) point scale
  Units on a Scale | 3.06 (1.09) | 3.14 (0.98) | 3.10 (1.02) | 3.25 (1.08) | 3.15 (1.05)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Daytime Nasal Symptoms Score
Description: Mean change from baseline in Daytime Nasal Symptoms score. Patients were asked to rate each of the 4 nasal symptoms of Congestion, Rhinorrhea, Itching, and Sneezing daily on a 4-point scale (0 (best) to 3 (worst)). The average of the 4 individual nasal symptoms scores was reported as the Daytime Nasal Symptoms Score.
Time Frame: Baseline and Week 2
Population: The primary efficacy analyses were based on the intention-to-treat (all-patients-treated) principle, i.e., all patients who had a baseline and at least one posttreatment measurement were included.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Montelukast | Loratadine | Montelukast/Loratadine
Number analyzed (Participants) | 148 | 151 | 300 | 298
Units on a Scale | -0.26 [-0.34 to -0.17] | -0.48 [-0.57 to -0.40] | -0.52 [-0.58 to -0.46] | -0.58 [-0.64 to -0.51]

2. Secondary Outcome: Mean Change From Baseline in Nighttime Symptoms Score
Description: Mean change from baseline in Nighttime Symptoms Score. Patients were asked to rate each symptom daily on a 4-point scale (0 (best) to 3 (worst)), and the combined score of Nasal Congestion Upon Awakening, Difficulty Going to Sleep, and Nighttime Awakenings was reported as the Nighttime Symptoms Score.
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Montelukast | Loratadine | Montelukast/Loratadine
Number analyzed (Participants) | 148 | 151 | 300 | 299
Units on a Scale | -0.12 [-0.20 to -0.04] | -0.29 [-0.37 to -0.22] | -0.26 [-0.31 to -0.20] | -0.28 [-0.34 to -0.23]

3. Secondary Outcome: Change From Baseline in Composite Symptoms Score (Daytime Nasal and Nighttime Symptoms)
Description: Composite Symptoms scores were computed as the average of the Daytime Nasal Symptoms scores and Nighttime Symptoms scores collected on a 4 point scale (0 (best) to 3 (worst)).
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Montelukast | Loratadine | Montelukast/Loratadine
Number analyzed (Participants) | 148 | 152 | 300 | 300
Units on a Scale | -0.2 [-0.28 to -0.12] | -0.40 [-0.48 to -0.33] | -0.41 [-0.47 to -0.35] | -0.45 [-0.50 to -0.39]

4. Secondary Outcome: Mean Change From Baseline in Daytime Eye Symptoms Score
Description: Mean change from baseline in Daytime Eye Symptoms scores. Patients were asked to rate each of the 4 eye symptom of tearing, itchy, red, and puffy eyes daily on a 4-point scale (0 (best) to 3 (worst)). The average of the 4 individual eye symptoms scores was reported as the Daytime Eye Symptoms Score.
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Montelukast | Loratadine | Montelukast/Loratadine
Number analyzed (Participants) | 148 | 151 | 299 | 298
Units on a Scale | -0.14 [-0.23 to -0.06] | -0.35 [-0.43 to -0.26] | -0.38 [-0.44 to -0.23] | -0.41 [-0.47 to -0.35]

5. Secondary Outcome: Mean Change From Baseline in Daytime Nasal Congestion Score
Description: Patients were asked to rate the nasal symptom of Congestion daily on a 4-point scale (0 (best) to 3 (worst)).
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Montelukast | Loratadine | Montelukast/Loratadine
Number analyzed (Participants) | 148 | 151 | 300 | 298
Units on a Scale | -0.19 [-0.29 to -0.09] | -0.41 [-0.51 to -0.31] | -0.39 [-0.46 to -0.32] | -0.43 [-0.50 to -0.36]

6. Secondary Outcome: Mean Change From Baseline in Daytime Rhinorrhea Score
Description: Patients were asked to rate the nasal symptom of Rhinorrhea daily on a 4-point scale (0 (best) to 3 (worst)).
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Montelukast | Loratadine | Montelukast/Loratadine
Number analyzed (Participants) | 148 | 151 | 300 | 298
Units on a Scale | -0.25 [-0.36 to -0.15] | -0.53 [-0.64 to -0.43] | -0.51 [-0.58 to -0.43] | -0.59 [-0.67 to -0.52]

7. Secondary Outcome: Mean Change From Baseline in Daytime Nasal Itching Score
Description: Patients were asked to rate the nasal symptom of Nasal Itching daily on a 4-point scale (0 (best) to 3 (worst)).
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Montelukast | Loratadine | Montelukast/Loratadine
Number analyzed (Participants) | 148 | 151 | 300 | 298
Units on a Scale | -0.26 [-0.37 to -0.16] | -0.49 [-0.60 to -0.39] | -0.56 [-0.64 to -0.48] | -0.62 [-0.70 to -0.55]

8. Secondary Outcome: Mean Change From Baseline in Daytime Sneezing Score
Description: Patients were asked to rate the nasal symptom of Sneezing daily on a 4-point scale (0 (best) to 3 (worst)).
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Montelukast | Loratadine | Montelukast/Loratadine
Number analyzed (Participants) | 133 | 138 | 278 | 272
Units on a Scale | -0.26 [-0.36 to -0.15] | -0.46 [-0.57 to -0.36] | -0.59 [-0.66 to -0.51] | -0.67 [-0.75 to -0.59]

9. Secondary Outcome: Mean Change From Baseline in Nasal Congestion Upon Awakening
Description: Patients were asked to rate the symptom of Nasal Congestion Upon Awakening daily on a 4-point scale (0 (best) to 3 (worst)).
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Montelukast | Loratadine | Montelukast/Loratadine
Number analyzed (Participants) | 148 | 151 | 300 | 299
Units on a Scale | -0.15 [-0.25 to -0.06] | -0.35 [-0.44 to -0.25] | -0.30 [-0.37 to -0.23] | -0.32 [-0.39 to -0.25]

10. Secondary Outcome: Patient's Global Evaluation of Allergic Rhinitis
Description: An evaluation by the patient, administered at the last visit (or upon discontinuation) using a 7-point scale, of the change in symptoms as compared to the beginning of the study. Responses were assigned numerical values from 0 (very much better) to 6 (very much worse).
Time Frame: Week 2
Population: The primary efficacy analyses were based on the intention-to-treat (all-patients-treated) principle. Since only 1 measurement was obtained during the treatment period, no missing values were imputed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Montelukast | Loratadine | Montelukast/Loratadine
Number analyzed (Participants) | 148 | 153 | 298 | 298
Units on a Scale | 2.37 [2.13 to 2.61] | 2.10 [1.86 to 2.33] | 2.00 [1.83 to 2.17] | 1.92 [1.74 to 2.09]

11. Secondary Outcome: Physician's Global Evaluation of Allergic Rhinitis
Description: An evaluation by the physician, administered at the last visit (or upon discontinuation) using a 7-point scale, of the change in symptoms as compared to the beginning of the study. Responses were assigned numerical values from 0 (very much better) to 6 (very much worse).
Time Frame: Week 2
Population: as for outcome 10
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Montelukast | Loratadine | Montelukast/Loratadine
Number analyzed (Participants) | 147 | 153 | 299 | 299
Units on a Scale | 2.35 [2.15 to 2.56] | 2.13 [1.93 to 2.33] | 2.05 [1.90 to 2.19] | 1.99 [1.84 to 2.13]

12. Secondary Outcome: Mean Change From Baseline in Rhinoconjunctivitis Quality-of-Life Score
Description: Patients completed a Rhinoconjunctivitis Quality-of-Life Questionnaire, 28 questions on a 7-point scale [0(best) to 6(worst)] across 7 domains: activities, sleep, non-nose/eye symptoms, practical problems, nasal symptoms, eye symptoms, emotional. Scores per domain were averaged, then scores for the 7 domains were averaged for an overall score.
Time Frame: Week 2
Population: The primary efficacy analyses were based on the intention-to-treat (all-patients-treated) principle, i.e., all patients who had a baseline and at least one posttreatment measurement were included. No missing values were imputed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Montelukast | Loratadine | Montelukast/Loratadine
Number analyzed (Participants) | 147 | 153 | 298 | 299
Units on a Scale | -0.80 [-0.98 to -0.63] | -1.09 [-1.26 to -0.92] | -1.06 [-1.19 to -0.93] | -1.16 [-1.29 to -1.03]

ADVERSE EVENTS:
Time Frame: During the 2 week, double-blind treatment period, and up to and including 14 days after the last dose of study therapy.
Description: Although a patient may have had two or more adverse experiences the patient is counted only once in a category. The same patient may appear in different categories.
Arm/Group | Placebo | Montelukast | Loratadine | Montelukast/Loratadine
Serious Adverse Events (participants affected / at risk) | 1/149 | 0/155 | 0/301 | 0/302
Other Adverse Events (participants affected / at risk) | 8/149 | 5/155 | 13/301 | 10/302
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=149) | Montelukast (N=155) | Loratadine (N=301) | Montelukast/Loratadine (N=302)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 — Pregnancies are not considered serious adverse events, however, they are collected in a similar manner so that they are learned of quickly and are followed to outcome. Therefore they appear as an event in our SAE reporting tables.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=149) | Montelukast (N=155) | Loratadine (N=301) | Montelukast/Loratadine (N=302)
Headache (Nervous system disorders) | 8 | 5 | 13 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.